CLINICAL TRIAL: NCT04361643
Title: Double-blind Randomized Controlled Clinical Trial of Low-dose Lenalidomide in the Treatment of COVID-19 Disease
Brief Title: Low-dose Lenalidomide for Non-severe COVID-19 Treatment Trial
Acronym: GETAFE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVID19-EC01
Record Dates: First submitted 2020-04-23; First posted 2020-04-24 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Patients will receive Lenalidomide as a 5 mg capsule PO daily, days 1, 3, and 5.
  Interventions: Drug: Lenalidomide as a 5 mg capsule PO daily, days 1, 3, and 5.
- Placebo (Placebo Comparator): Patients will receive a placebo capsule PO daily, days 1, 3, and 5.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lenalidomide as a 5 mg capsule PO daily, days 1, 3, and 5. — Patients will receive Lenalidomide as a 5 mg capsule PO daily, days 1, 3 and 5, together with a prophylactic dose of low molecular weight heparin (LMWH) or therapeutic dose if needed due to previous comorbidity.
  Other Names: Revlimid
  Arms: Experimental
Drug: Placebo — Patients will receive a placebo capsule PO daily, days 1, 3 and 5, together with a prophylactic dose of low molecular weight heparin (LMWH) or therapeutic dose if needed due to previous comorbidity.
  Arms: Placebo

SUMMARY:
Double-blind randomized controlled clinical trial (RCT) of low-dose lenalidomide in the treatment of elderly patients (> 60 years of age) with mild to moderate clinical signs of COVID-19 disease from the Hospital Universitario of Getafe.

The study will include patients of both sexes (> 60 years of age) with mild to moderate clinical presentation of COVID-19 (ROX index > 10). Subjects will be randomly assigned to the experimental arm with lenalidomide (5 mg/24h, day 1, 3 and 5) or to the controlled arm. Other concomitant medication for the treatment of COVID-19 will be also considered.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 60 years of age
* Diagnosed case (PCR test for COVID-19 if available) or COVID-19 clinical symptoms (defined as fever, dry cough, dyspnea, chest radiography with compatible findings with COVID-19)
* Lymphocyte count ≥ 0.2 x 103/µL and ≤1.0 x 103/µL.
* Neutrophil count ≥ 1.8 x 103/µL, platelets ≥ 150 x 103/µL.
* ROX ≥ 10 index
* Signed informed consent document
* Willing to comply with the lenalidomide Risk Minimization Program (Pregnancy Prevention Program approved)

Exclusion Criteria:

* Absolute contraindication of lenalidomide use or hypersensitivity to the active ingredient or any of the excipients.
* Active neoplasia
* Previous autoimmune disease
* Concurrent infection of HBV, HCV or tuberculosis.
* Aspartate transaminase (AST) or alanine transaminase (ALT) > 3 times the upper limit of normal (ULN).
* Bilirubin levels > 1.5 times the ULN
* Renal impairment with an estimated GF < 30ml/min
* Venous thromboembolism events within the previous 3 years
* Significant active heart disease within the previous 6 months, including congestive heart failure (class II-IV NYHA), unstable angina or myocardial infarctions
* Sexually active subjects who refuse the lenalidomide Risk Minimization Program
* Inability to comply with the working protocol under the responsible health professional opinion.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-27 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 30 days
  Days to clinical recovery or days until discharge
Immune-inflammatory improvement | 30 days
  o Improvement of the neutrophil-to-lymphocyte ratio (NLR)

SECONDARY OUTCOMES:
Mortality | 30 days
  All-cause mortality at 30 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin De Haro, MD, Study Chair — Hospital Universitario Getafe
Locations (1):
- Hospital Universitario de Getafe, Getafe, Spain

IPD SHARING:
Plan to Share IPD: No